CLINICAL TRIAL: NCT03122132
Title: Efficacy and Safety in Clinical Practice of Ombitasvir/Paritaprevir/ Ritonavir and Dasabuvir Administered for 8 Weeks (3D8) in Treatment-naïve Genotype 1b Hepatitis C Virus Infected Patients: Analysis of Data From Hepa-C Registry.
Brief Title: Effectiveness, Safety and Clinical Outcomes of Paritaprevir/Ombitasvir/r+Dasabuvir 8 Weeks
Acronym: 3D8
Status: Completed | Type: Observational
Sponsor: Hepa C (Other)
Responsible Party: Sponsor
Other Study IDs: 0002
Record Dates: First submitted 2017-04-11; First posted 2017-04-20 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Hepatitis C Infection
Keywords: Hepatitis C Infection; Ombitasvir/Paritaprevir/Ritonavir+dasabuvir
MeSH Terms: conditions — Hepatitis C | interventions — ombitasvir; paritaprevir; Ritonavir; dasabuvir

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spanish cohort with HCV treated with DAA: Spanish cohort with HCV treated in real practice with ombitasvir/paritaprevir/ritonavir 8 weeks and dasabuvir 8 weeks
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir 8 weeks; Drug: dasabuvir 8 weeks

INTERVENTIONS:
Drug: ombitasvir/paritaprevir/ritonavir 8 weeks — Spanish cohort with HCV treated in real practice with ombitasvir/paritaprevir/ ritonavir 8 weeks
  Other Names: viekirax
Drug: dasabuvir 8 weeks — Spanish cohort with HCV treated in real practice with dasabuvir 8 weeks
  Other Names: exviera

SUMMARY:
The aim of the study is to evaluate in clinical practice the efficacy and safety of ombitasvir/paritaprevir/ ritonavir and dasabuvir administered for 8 weeks in treatment-naïve participants with genotype 1b hepatitis C virus (HCV).

DETAILED DESCRIPTION:
HCV chronic infection affects 200 million people worldwide. HCV antiviral treatment has evolved rapidly since 2011. The introduction of direct-acting antivirals (DAAs) achieve great effectiveness with minimum SAEs and short treatment duration. However, studies evaluating efficacy and safety of ombitasvir/paritaprevir/ ritonavir and dasabuvir during 8 weeks are limited in real clinical practice. The aim of the study is to evaluate in clinical practice the efficacy and safety of ombitasvir/paritaprevir/ ritonavir and dasabuvir administered for 8 weeks in treatment-naïve participants with genotype 1b hepatitis C virus (HCV).

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C (anti-HCV antibodies and detectable HCV-RNA).
* Genotype 1b infection
* Treatment-naïve and non-cirrhotic

Exclusion Criteria:

* HCV genotype or subtype other than GT1b.
* Any current or past clinical evidence of cirrhosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HCV who are treated in real practice with Ombitasvir/Paritaprevir/Ritonavir+Dasabuvir
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Sustained virological response 12 weeks post-treatment (SVR12) | 12 weeks after the last dose of study drug
  Percentage of participants who achieve sustained virological response 12 weeks post-treatment (SVR12)
  • Measure: Hepatitis C virus ribonucleic acid (HCV-RNA) levels less than the lower limit of quantification.

SECONDARY OUTCOMES:
Percentage of patients with virologic failure during treatment | Up to 12 weeks after last dose of study drug
  Percentage of patients with virologic failure during treatment
  • Measure: Percentage of patients with confirmed >=1 log10 IU/mL increase from nadir in HCV RNA at any time point during treatment
Mild fibrosis and sustained virological response 12 weeks post-treatment | Up to 12 weeks after last dose of study drug
  Percentage of patients with mild fibrosis who achieve sustained virological response 12 (SVR12) weeks post-treatment
  • Measure: percentage of patients with a baseline transient elastography < 6 kPa
Percentage of participants with low baseline viral load and SVR12 weeks post-treatment | Baseline and 12 weeks after the last dose of drug
  Percentage of participants with low baseline viral load who achieve sustained virological response 12 (SVR12) weeks post-treatment
  • Measure: HCV RNA levels less than the lower limit of quantification.

CONTACTS AND LOCATIONS:
Locations (1):
- Carrion, Jose Antonio, PhD, Barcelona, Spain

REFERENCES:
- [Derived] Puigvehi M, De Cuenca B, Viu A, Diago M, Turnes J, Gea F, Pascasio JM, Lens S, Cabezas J, Badia E, Olveira A, Morillas RM, Torras X, Montoliu S, Cordero P, Castro JL, Salmeron J, Molina E, Sanchez-Ruano JJ, Moreno J, Anton MD, Moreno JM, De la Vega J, Calleja JL, Carrion JA. Eight weeks of Paritaprevir/r/Ombitasvir + Dasabuvir in HCV genotype 1b with mild-moderate fibrosis: Results from a real-world cohort. Liver Int. 2019 Jan;39(1):90-97. doi: 10.1111/liv.13950. Epub 2018 Nov 12. PMID 30160363